CLINICAL TRIAL: NCT06951386
Title: The Impact of 12 Weeks Intervention With Plant-based Oat Drink Rich in Short-chain Fatty Acids on Postprandial Lipidemia in Individuals at Risk for Metabolic Syndrome
Brief Title: The Impact of Daily Intake of Short-chain Fatty Acids on Cardiometabolic Risk Factors in Individuals at Risk for Metabolic Syndrome
Acronym: 12OATS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Prof., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: S69712
Record Dates: First submitted 2025-01-29; First posted 2025-04-30 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-01

CONDITIONS: Energy Expenditure; Metabolic Syndrome; Anthropometry; Body Composition; Glycemia; Lipaemia; Metabolomics; Blood Pressure
Keywords: short-chain fatty acids; cardiometabolic health
MeSH Terms: conditions — Metabolic Syndrome; Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drink enriched with short-chain fatty acids (Active Comparator): Treatment with enriched drink
  Interventions: Dietary Supplement: with short-chain fatty acids enriched drink
- Control drink (Placebo Comparator): Treatment with control drink
  Interventions: Dietary Supplement: unenriched oat drink

INTERVENTIONS:
Dietary Supplement: with short-chain fatty acids enriched drink — Oat-based drink enriched with 15 g/L short-chain fatty acids
  Arms: Drink enriched with short-chain fatty acids
Dietary Supplement: unenriched oat drink — Oat-based drink
  Arms: Control drink

SUMMARY:
During this study, the effect of short-chain fatty acids on blood lipaedemia, glycemia, anthropometrics, blood pressure and energy expenditure will be investigated.

DETAILED DESCRIPTION:
The goal of this study is to investigate the impact of consuming every day a drink enriched with short-chain fatty acids for 12 weeks on the cardiometabolic health in individuals at risk of metabolic syndrome. This means the investigators are looking for people with overweight and disrupted cholesterol, high blood pressure or elevated blood glucose. The individuals will consume for 12 weeks a drink either enriched with SCFA or a control drink (randomly allocated). Before and after this period (study visit 1 and 4), a study visit will take place in which metabolic parameters will be measured such as blood pressure, body weight, waist- and hip circumference, body composition, energy expenditure, glucose, insulin and blood lipids. After 4 and 8 weeks, anthropometrics, blood pressure and body composition will be measured during a short study visit (study visit 2 and 3).

ELIGIBILITY:
Inclusion Criteria:

* male and female participants
* central obesity ( BMI ≥ 25 kg/m² or waist circumference ≥ 80 cm for women/ ≥ 94 cm for men)
* One additional risk factor for metabolic syndrome:

  1. Insulin resistance (HOMA-IR ≥ 1.7 or fasting glucose ≥ 100 mg/dl)
  2. Triglyceride concentration ≥ 150 mg/dl
  3. HDL-cholesterol < 40 mg/dl for women/ < 50 mg/dl for men
  4. Systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥ 85 mmHg
* knowledge of English

Exclusion Criteria:

* gastrointestinal disorders such as IBD, IBS, celiac disease, chronic constipation, chronic diarrhoea
* history of abdominal surgery, except for appendectomy
* Use of antihypertensive, cholesterol lowering, glucose-regulating drugs and corticosteroids
* Use of antibiotics 3 months prior to the start or during the study
* Use of probiotics and prebiotics 2 weeks prior to the start of the study/ during the study
* Being on weight loss, gluten-free, lactose-free or vegan diet
* Pregnancy, lactation or wish to become pregnant
* Previous or current substance/ alcohol dependence or abuse
* Hyper- or hypothyroidism
* Allergy or intolerance to oat milk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Fasting triglycerides | During study visit 1(baseline) and visit 4 (end of intervention, week 12)
  Triglyceride concentrations will be measured in fasting state

SECONDARY OUTCOMES:
Fasting glycemia | During study visit 1 (baseline) and 4 (12 weeks)
  In fasting state glucose will be measured
Fasting energy expenditure | During study visit 1 (baseline) and 4 (12 weeks)
  Energy expenditure will be measured for 30 minutes in fasting state using indirect calorimetry
Anthropometrics: body weight | Baseline, week 4, week 8 and week 12
  Body weight will be measured at the start of the visit
Blood pressure | Baseline, week 4, week 8 and week 12
  Systolic and diastolic blood pressure will be measured at the start of the visit
Insulin resistance: HOMA-IR | During study visit 1 (baseline) and 4 (12 weeks)
  HOMA-IR will be determined using fasting and postprandial (after 30 min) glucose and insulin levels.
HbA1c | During study visit 1 (baseline) and 4 (12 weeks)
  Glycosylated hemoglobin HbA1c will be measured in fasting state
Short-chain fatty acids in stool | Within 2 days prior to study visit 1 (baseline) and 4 (12 weeks)
  Short-chain fatty acids in stool will be measured before and after the intervention
Incretin hormone GLP1 | During study visit 1 (baseline) and 4 (12 weeks) (up to 6 hours)
  GLP-1 will be measured in fasting and postprandial state (30, 60, 90, 120, 150,180, 240, 300, 360 min)
Cytokines | During study visit 1 (baseline) and 4 (12 weeks)
  Cytokines such as IL-1β, IL-6, IL-10, TNF-alpha, IL-13 and interferon (IFN)-γ will be measured in fasting state (unit: pg/ml)
24 hour diet recall | Before the intervention and during week 4, 8 and 12 of the intervention
  Subjects will complete an online 24 hour diet recall
Postprandial glycemia | During study visit 1 (baseline) and 4 (12 weeks) (up to 6 hours)
  Glucose concentrations will be measured 30,60,90,120,150,180,240,300 and 360 min after a mixed meal tolerance test
Postprandial lipaedemia: triglycerides | During study visit 1 (baseline) and 4 (12 weeks) (up to 6 hours)
  Triglycerides will be measured after a mixed meal tolerance test (30, 60, 90, 120, 150, 180, 240, 300, 360 min)
Short-chain fatty acids in blood | During study visit 1 (baseline) and 4 (12 weeks) (up to 6 hours)
  Short-chain fatty acids (acetate, propionate and butyrate) concentrations will be measured in fasting and postprandial state (30, 60, 90, 120, 180, 240, 300, 360 min).
Appetite measurements | During study visit 1 (baseline) and 4 (12 weeks) (up to 6 hours)
  Appetite in response to mixed meal tolerance test, will be measured using 100 millimeter (mm) Visual Analogue Scale (indicating score on line of 100 mm, 0 mm: don't agree, 100 mm: totally agree) in fasting (i.e. 0 minute) and postprandial state (30, 60, 90, 120,150, 180, 240, 300 and 360 min).
Physical activity measurement | At the end of study visit 1 (baseline) and 4 (12 weeks)
  Individuals complete the short form of the international physical activity questionnaire (IPAQ) before and after the intervention. In the IPAQ participants fill in the number of days/ week they spent doing vigorous, moderate activity and walking and how long (hours and minutes) per day they do this. It also includes a question about how long they sit on a day.
Postprandial energy expenditure | During study visit 1 (baseline) and 4 (12 weeks) (up to 3 hours)
  Energy expenditure will be measured for 3 hours after the mixed meal tolerance test
Fasting blood lipids | During study visit 1 (baseline) and 4 (12 weeks)
  Total, HDL-, LDL-cholesterol (mg/dl) will be measured in fasting state
Metabolomics | During study visit 1 (baseline) and 4 (12 weeks)
  Untargeted metabolomics analysis will be performed on fasting blood sample
Fasting insulinemic response | During study visit 1 (baseline) and 4 (12 weeks)
  In fasting state the insulin concentration will be measured
Anthropometrics: waist and hip circumference | Baseline, week 4, week 8 and week 12
  Waist- and hip circumference will be measured at the start of the visit
Gut hormone: PYY | During study visit 1 (baseline) and 4 (12 weeks) (up to 6 hours)
  PYY will be measured in postprandial state at 30, 60, 90, 120, 180, 240, 300 and 360 min
LBP | During study visit 1 (baseline) and 4 (12 weeks)
  LBP will be measured in fasting state
HOMA-B | During study visit 1 (baseline) and 4 (12 weeks)
  HOMA-B will be measured in fasting state
Insulinogenic index | During study visit 1 (baseline) and 4 (12 weeks)
  IGI will be measured in fasting state. IGI is ratio of (postprandial insulin (30 min) -fasting insulin (mU/L)) over (postprandial glucose (30 min) - fasting glucose (mmol/L))
Postprandial insulin | During study visit 1 (baseline) and 4 (12 weeks) (up to 6 hours)
  Insulin concentrations will be measured 30,60,90,120,150,180,240,300 and 360 min after a mixed meal tolerance test
Postprandial lipaedemia: total, LDL and HDL cholesterol | During study 1 (baseline) and study 4 (12 weeks) (up to 6 hours)
  Total, HDL and LDL cholesterol will be measured after 30,60,90,120,150,180,240,300 and 360 min (mg/dl)
Postprandial lipaedemia: free fatty acids | During study 1 (baseline) and study 4 (12 weeks) (up to 6 hours)
  Free fatty acids will be measured at 30,60,90,120,150,180,240,300 and 360 min (µmol/l)
% fat mass | During all 4 study visits (0, 4,8 and 12 weeks) (fasted state)
  % fat mass is measured using a bodystat bioelectrical impedance device, expressed in %
kg fat mass | During all 4 study visits (0, 4,8 and 12 weeks) (fasted state)
  kg fat mass is measured using a bodystat bioelectrical impedance device, expressed in kg
fat free mass (kg) | During all 4 study visits (0, 4,8 and 12 weeks) (fasted state)
  Fat free mass is measured using a bodystat bioelectrical impedance device, expressed in kg
Dry lean weight (kg) | During all 4 study visits (0, 4,8 and 12 weeks) (fasted state)
  Dry lean weight is measured using a bodystat bioelectrical impedance device, expressed in kg
Water percentage | During all 4 study visits (0, 4,8 and 12 weeks) (fasted state)
  % water in body is measured using a bodystat bioelectrical impedance device, expressed in %
Total body water (L) | During all 4 study visits (0, 4,8 and 12 weeks) (fasted state)
  Volume of body water is measured using a bodystat bioelectrical impedance device, expressed in liters
Average energy requirements | During all 4 study visits (0, 4,8 and 12 weeks) (fasted state)
  Average energy requirements is measured using a bodystat bioelectrical impedance device, expressed in kcal/day
Basal metabolic rate | During all 4 study visits (0, 4,8 and 12 weeks) (fasted state)
  Basal metabolic rate (BMR) is measured using a bodystat bioelectrical impedance device, expressed in kcal/day
basal metabolic rate (BMR)/ body weight | During all 4 study visits (0, 4,8 and 12 weeks) (fasted state)
  BMR/body weight is measured using a bodystat bioelectrical impedance device, expressed in kcal/kg
BMI | During all 4 study visits (0, 4,8 and 12 weeks) (fasted state)
  BMI is measured using a bodystat bioelectrical impedance device, expressed in kg/m²
Waist to hip ratio | During all 4 study visits (0, 4,8 and 12 weeks) (fasted state)
  Waist to hip ratio is measured using a bodystat bioelectrical impedance device
Resistance during bioelectrical impedance | During all 4 study visits (0, 4,8 and 12 weeks) (fasted state)
  Resistance is measured using a bodystat bioelectrical impedance device, expressed in Ohm
Free fatty acids in fasting state | During study visit 1 (baseline) and 4 (after 12 weeks)
  Free fatty acids will be measured in fasted state (µmol/l)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Verbeke, Prof., Principal Investigator — KU Leuven
Locations (1):
- KU Leuven/ UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
No IPD data will be shared with other researchers.